CLINICAL TRIAL: NCT06159686
Title: This Study Aims to Compare the Efficacy of Hemp-containing Cream and a Placebo in the Treatment of Uremic Pruritus in Hemodialysis Patients. Patients Were Randomly Assigned Either the Hemp-containing Cream or a Placebo and Evaluated the WI-NRS and Skindex-10 Scores at Week 2, 4.
Brief Title: The Efficacy of Hemp-containing Cream Versus Placebo in the Treatment of Uremic Pruritus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Suthiya Anumas, Principal Investigator, Thammasat University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 074/2566
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Uremic Pruritus
Keywords: Hemp; Uremic pruritus; hemodialysis; cannabinoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hemp group (Experimental): They was assigned to apply the hemp-containing cream.
  Interventions: Drug: Hemp
- Control group (Placebo Comparator): They was assigned to apply the placebo cream.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hemp — The application of the hemp-containing cream occurred in the morning and evening on the itching areas, excluding the face for 4 weeks.
  Arms: hemp group
Drug: Placebo — The application of the placebo cream occurred in the morning and evening on the itching areas, excluding the face for 4 weeks.
  Arms: Control group

SUMMARY:
Uremic pruritus is a significant burden on hemodialysis patients, affecting approximately 46% of individuals undergoing dialysis. Various mechanisms, including inadequate dialysis, increased uremic toxins, inflammatory cytokines, parathyroid hormone, phosphorus, dry skin, mast cell histamine secretion, and nerve stimulation through μ-opioid receptors and nociceptors, contribute to uremic pruritus. Current treatments include antihistamines, gabapentin, moisturizer creams, and capsaicin creams, with limited success, as only 10% of patients find relief. Cannabinoids were also mentioned in uremic pruritus treatment but are less commonly used and there are no randomised controlled trial. Cannabinoid binding to CB1 and CB2 receptors inhibits mast cell differentiation, aggregation, and histamine release, whereas cannabinoid binding to TRP-iron receptors reduces peripheral nerve activation. Thus, cannabinoid seem to effective in relieving pruritus via various mechanisms.

This study aims to assess the effectiveness of a hemp-containing cream in comparison to a placebo for treating uremic pruritus among hemodialysis patients.

DETAILED DESCRIPTION:
Eligible participants is randomly assigned in a 1:1 ratio to receive either a hemp-containing cream or a placebo. then, they are assessed for the severity of itching symptoms using the WI-NRS and their itch-related quality of life using the Skindex-10 score at baseline, week 2, and week 4 of the study. Additionally, adverse effects are documented. Data is collected by the research assistant and recorded in computer with locking password and also was validated with second assistant.

We planned for a sample size of 60 participants to detect differences in itchinEligible participants is randomly assigned in a 1:1 ratio to receive either a hemp-containing cream or a placebo. then, they are assessed for the severity of itching symptoms using the WI-NRS and their itch-related quality of life using the Skindex-10 score at baseline, week 2, and week 4 of the study. Additionally, adverse effects are documented. Data is collected by the research assistant and recorded in computer with locking password and also is validated with second assistant.

For statistical analysis, continuous variables are compared using an unpaired t-test or Mann-Whitney U test, as appropriate. Categorical variables are compared using a Chi-square test or Fisher's exact test. The adjusted mean difference is used Analysis of Covariance (ANCOVA) , adjusted by score at baseline.

All statistical analyses were performed using Stata v.17.0 (StataCorp, Texas).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old, diagnosed with end-stage kidney disease
* Undergoing thrice-weekly chronic hemodialysis for more than 90 days
* Exhibit a WI-NRS score of 3 or higher

Exclusion Criteria:

* Ahistory of hemp allergy
* Pregnancy or breastfeeding
* Dermatologic diseases
* Adjustments to medications for controlling itch within the 14 days preceding the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
WI-NRS (Worst Itching Numerical Rating scale) score at week 4 | week 4
  WI-NRS score will demonstrate the severity of itch at week 4. The minimum score is 0 and maximum score is 10. The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
WI-NRS at week 2 | week 2
  WI-NRS score will demonstrate the severity of itch at week 2. The minimum score is 0 and maximum score is 10. The higher scores mean a worse outcome. The minimum score is 10 and maximum score is 60. The higher scores mean a worse outcome.
Skindex-10 score at weeks 2 and 4 | week 2 and 4
  Skindex-10 score will demonstrate the itch-related quality of life at week 2 and 4. The minimum score is 10 and maximum score is 60. The higher scores mean a worse outcome.
the mean difference score between baseline and week 4 for WI-NRS and the Skindex-10 score | week 4
  The change of WI-NRS score and Skindex-10 score between baseline and week 4 represents the change of severity and QOL after complete study (week4) compare to baseline. The greater different scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Suthiya Anumas, Principal Investigator — Thammasat University
Locations (1):
- Thammasat, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anumas S, Kuropakornpong P, Chakkavittumrong P, Tasanarong A, Pattharanitima P. Cannabis-Containing Cream for CKD-Associated Pruritus: A Double-Blind, Placebo Controlled Trial. Kidney Med. 2024 Aug 21;6(10):100894. doi: 10.1016/j.xkme.2024.100894. eCollection 2024 Oct. PMID 39328960